CLINICAL TRIAL: NCT02087384
Title: Quadrivalent HPV Vaccination After Effective Treatment of Anal Intraepithelial Neoplasia in HIV+ Men
Brief Title: HPV (Human Papilloma Virus) Vaccination After Treatment of Anal Intraepithelial Neoplasia (AIN)
Acronym: VACCAIN-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Jan Prins (Other)
Responsible Party: Sponsor-Investigator, Prof. Jan Prins, Professor. dr. J.M. Prins, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL45200.018.13
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: AIN; HIV
Keywords: Anal intraepithelial neoplasia; HIV; HPV; Vaccination; Gardasil; Prophylactic
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gardasil (Experimental): Gardasil
  Interventions: Biological: Gardasil
- Placebo (Placebo Comparator): Intramuscular Saline 0.9% vaccination at 0, 2 and 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Gardasil — Intramuscular Gardasil vaccination at 0, 2 and 6 months.
  Other Names: Quadrivalent HPV vaccine; Vaccine against HPV-6, 11, 16, 18
  Arms: Gardasil
Drug: Placebo — injection of 0.9% saline
  Other Names: intramuscular Saline 0.9%
  Arms: Placebo

SUMMARY:
This study evaluates vaccination with the quadrivalent HPV vaccine (Gardasil) versus placebo vaccination on prevention of high grade AIN recurrence in HIV-positive MSM (men who have sex with men) who were successfully treated for high grade AIN.

DETAILED DESCRIPTION:
Rationale: Since the introduction of combination antiretroviral therapy (cART), human immunodeficiency virus (HIV)-related morbidity and mortality have considerably decreased. However, as a result of the significantly prolonged life span, new causes of morbidity and mortality have become evident. In particular, anal cancer incidence has increased dramatically in HIV-positive men. Like cervical cancer, anal cancer is causally linked to infections with high-risk papillomaviruses, and is preceded by precursor lesions: anal intraepithelial neoplasia (AIN). Over 90% of HIV-positive MSM (men who have sex with men) have persisting anal HPV (human papilloma virus) infection, and high-grade (HG) AIN is present in 30% of all HIV+ MSM.

As in cervical intraepithelial neoplasia, early diagnosis and treatment of AIN have been advocated to prevent malignancy. Electrocoagulation/ cauterization is standard of care for intra-anal AIN, but after treatment, recurrence of lesions occurs in approx. 50% of cases. This is a major problem in an effective screening program for AIN.

In a nonconcurrent, non-blinded cohort study qHPV (quadrivalent human papilloma virus) vaccination significantly (HR 0.50) reduced HG AIN recurrence among MSM successfully treated for AIN. This is in accordance with findings in women treated for cervical intraepithelial neoplasia. Previous vaccination with quadrivalent HPV vaccine among women who had surgical treatment for HPV related disease significantly reduced the incidence of subsequent HPV related disease, including high grade disease.

Therefore, a strategy that is worth investigating is vaccination with the qHPV vaccine to prevent recurrences in HIV+ MSM who were successfully treated for HG AIN.

Objective: The primary objective of the current study is to assess the efficacy of qHPV vaccination in preventing recurrence of high-grade AIN in HIV+ MSM with CD4 counts >350 x 10E6/l who were successfully treated for high-grade intra-anal AIN in the past year.

Study population: HIV-positive MSM with a CD4 count > 350 cells/ul and intra-anal high-grade AIN (grade 2-3) that was successfully treated in the past year with conventional cauterization, cryotherapy, or other forms of local treatment.

Study design: A multicenter, randomised, double-blind clinical trial in four hospitals in the Netherlands.

Intervention: Patients are randomised for vaccination with the quadrivalent HPV vaccine (Gardasil ®) or vaccination with a matching placebo at months 0, 2 and 6.

Randomisation will be stratified for complete response versus partial response (from HG AIN to low-grade (LG) AIN) of the initial HG AIN lesion, for treatment less than 6 months ago versus treatment 6 months and longer ago, and for AMC versus other hospitals.

Main study parameters/endpoints: Screening for AIN will be performed by high-resolution anoscopy (HRA), at inclusion (first vaccination) and at last vaccination (6 months), and repeated at 6 and 12 months after the last vaccination. Safety Monitoring for adverse events and injection-site reactions will be performed one week after each vaccination and thereafter every 6 months for a total of 12 months of follow-up.

Primary end point will be the cumulative recurrence of HG AIN at 12 months after the last vaccination, as assessed by HRA (High-Resolution Anoscopy), with biopsies taken of suspect lesions.

Secondary outcome measures are toxicity/ safety, recurrence of HG AIN at last vaccination and 6 months afterwards, cumulative occurrence of LG AIN at 12 months after the last vaccination, cumulative occurrence of anogenital warts at 12 months after the last vaccination, causative HPV type in recurrent AIN lesions, as assessed by LCM (Laser Capture Microdissection)/ PCR (polymerase chain reaction), and HPV type-specific antibody response.

The total sample size is estimated to be 125 patients based on an expected recurrence rate of 50% within 12 months. Statistical analysis will be based on the intention-to-treat principle. Both primary and secondary endpoints will be analyzed by descriptive statistics and the chi-square test with a 0,05 two-sided significance level.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

HIV+ MSM who were successfully treated for HG AIN are still at a 50% risk for recurrences, with additional treatment sessions needed, and an ongoing risk for malignant degeneration of lesions.

Costs of 3 vaccinations are approx. € 400, but if vaccination reduces recurrence rates by 50%, this will be a highly cost-effective intervention, very likely to be introduced into regular care.

For the study, patients will be vaccinated 3 times with the quadrivalent vaccine Gardasil ® or placebo, and will undergo two extra HRAs. Clinical trial data show that the most common adverse events of Gardasil ® were mild or moderate, so few risks are associated with study participation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age ≥ 18 years.
* HIV+ MSM, CD4 count > 350/ul (maximum 6 months before screening visit).
* Biopsy-proven intra-anal high-grade AIN successfully treated in the past year with cauterization, cryotherapy, Efudix, imiquimod or another form of local treatment. A maximum interval of 1 year between last treatment and first vaccination is allowed. Lesions with regression from HG to LG AIN (AIN 1) will also be eligible.
* Lesions (still) in remission:

  * Remission has to be established by 2 independent HRA anoscopists.
  * A maximum interval of 3 months is allowed between the first of these HRAs and the first vaccination, and a maximum interval of 6 weeks is allowed between the second of these HRAs and the first vaccination.
  * Biopsies of suspect lesions need to be obtained in one of the HRA sessions.
* Good performance status (a Karnofsky performance score of ≥ 60 [on a scale of 0 to 100, with higher scores indicating better performance status]).
* Pre-treatment haematology, and plasma ASAT, ALAT and creatinine levels compatible with study inclusion (maximum 6 weeks before screening visit).

Exclusion criteria:

* Immunosuppressive medication or other diseases associated with immunodeficiency.
* Life expectancy less than one year.
* Previous HPV vaccination.
* History of anal cancer.
* Other diseases not compatible with study participation.
* Allergy against constituent of Gardasil ® vaccine.
* Currently peri-anal AIN2 or 3.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Cumulative recurrence of intra-anal or peri-anal HG AIN at 12 months after the last vaccination (18 months after inclusion), as assessed by HRA, with biopsies taken of suspect lesions. | 18 months

SECONDARY OUTCOMES:
Toxicity/ safety of the Gardasil vaccine in HIV+ MSM. | 18 months
  One week after each vaccination and during all follow up visits the most common adverse events of Gardasil and other eventually occuring complaints will be evaluated by history taking. Adverse events will be graded according to the CTCAE v4 (Common Terminology Criteria for Adverse Events), which grades events on a scale of 1 to 5, with higher grades indicating greater severity.
Recurrence of intra-anal or peri-anal HG AIN at the moment of last vaccination and 6 months afterwards. | 6 and 12 months
Cumulative occurrence of intra-anal or peri-anal LG AIN at 12 months after the last vaccination. | 18 months
  The patients with LG AIN at inclusion are excluded from this analysis.
Cumulative occurrence of anogenital warts at 12 months after the last vaccination. | 18 months
  Evaluated by physical examination and history taking.
Causative HPV type in recurrent AIN lesions, as assessed by LCM/ PCR. | 18 months
HPV type-specific antibody response. | 9 months (3 months after last vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, prof, MD, infectiologist, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Henry JC de Vries, prof, MD, dermatologist, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (3):
- Netherlands (3):
  - DC Klinieken Oud Zuid, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02087384/SAP_000.pdf